CLINICAL TRIAL: NCT00190008
Title: Therapeutic Use of Piracetam for Treatment of Patients Suffering From Tardive Dyskinesia: a Double Blind, Placebo-Controlled Crossover Study
Brief Title: Piracetam for Treatment Tardive Dyskinesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BMHC-3529
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Tardive Dyskinesia
Keywords: tardive dyskinesia; piracetam
MeSH Terms: conditions — Tardive Dyskinesia | interventions — Piracetam

INTERVENTIONS:
Drug: piracetam

SUMMARY:
The mechanism involved in the development of tardive dyskinesia (TD) is complicated. It now seems that several neurotransmitter systems may be affected, including dopaminergic, noradrenergic, gamma-amino-butyric acid (GABA) ergic, cholinergic and peptidergic pathways.

Piracetam (2-oxo-pyrrolidone) is a nootropic drug structurally related to GABA. It has been used clinically to treat a wide range of diseases and conditions, mainly in treatment of organic brain syndrome, myoclonus, memory impairment, post-concussional syndrome, vertigo, alcohol withdrawal, cerebrovascular insufficiency, hypoxia, intoxications of different origins or mechanic brain injures. Piracetam is cerebral homeostatic normalizer, neuroprotectant, cerebral metabolic enhancer and brain integrative agent. It enhances brain energy, especially under deficit condition: hypoxia, chemical toxicity or impaired cerebral microcirculation; preserve, protect and enhance synaptic membrane and receptor structure and plasticity. It has various effects on glutamate neurotransmission on micromolar levels piracetam potentiates potassium-induced release of glutamate from hippocampal nerves. It is an oxidant agent and may be useful for treatment TD. Piracetam is among the toxicologically safest drugs ever developed even in mega doses.

Data derived from some clinical reports have suggested that piracetam can improve symptoms and is effective agent for treatment of different movement disorders including acute neuroleptic induced extrapyramidal symptoms and TD. The doses that used for TD treatment varied from 800 mg/day to 24000 mg/day. According to these findings the symptoms of TD disappeared in the period of 3-7 days.

To date there was only one double-blind crossover study regarding use of piracetam for treatment TD that was conducted almost 20 years ago. The findings of this study were impressive, but to our knowledge nobody reproduced these results.

DETAILED DESCRIPTION:
We intend to examine 40 inpatients, aged 18-75 years old, suffering from TD and its variants. Criteria for inclusion into the study will be: a) DSM-IV diagnosis of tardive dyskinesia; b) stable psychotropic regimen of a month prior to entry into the study; c) duration of TD of at least 1 year; d) all patients had to be hospitalized.

Exclusion criteria will be: a) evidence of family history of Huntington's disease; b) evidence of substance or alcohol abuse; c) patients who received any form of vitamin medication; d) patients with concurrent medical illness or neurological disorders that may have influenced up the diagnosis of tardive dyskinesia.

The study design will be a double blind, randomized crossover group study and will be last for 8 weeks. This period provided an opportunity to exclude the influence of spontaneous fluctuations in the severity of TD. Full physical and laboratory examinations were performed on all inpatients in the beginning and at the end of the trial. Psychotropic medication will be maintained at fixed doses throughout the duration of study. The capsules preparations will be made by a professional pharmacist in the same size and color capsules in individual number-coded packages. The capsules will be added to the patients' usual medications and will be given by nurses.

Assessments for tardive dyskinesia and its variants will be done using Extrapyramidal Symptom Rating Scale (ESRS) at baseline and repeated every week, prior crossover, and then every week. This scale was developed by G. Chouinard and A. Ross-Chouinard (15) and was designed to rate three types of extrapyramidal symptoms: parkinsonian, dystonic and dyskinetic. Although the scale may be applied to non-drug-induced extrapyramidal symptoms, its sensitivity has been most often assessed in the evaluation of drug-induced extrapyramidal symptoms. The dose of piracetam or placebo will be increased every week on 2000 mg up to 8000 mg/day in dependence on the changes of movement disorders. The doses of their neuroleptic medications not will be change a month before and during the research. The patients will take piracetam or placebo as addition to their constant medication.

It should be emphasized again that improvement of TD symptoms after piracetam addition was appeared through very short period (3-7 days) in comparison to other medications used for treatment of TD. Moreover, if efficacy of piracetam will be proved in our study, clinicians obtain a new, effective, safe drug for TD treatment with rapid onset of the action.

References

1. Lohr JB. Oxygen radicals and neuropsychiatric illness. Some speculations. Arch Gen Psychiatry 1991;48(12):1097-1106.
2. Gouliaev AH, Senning A. Piracetam and other structurally related nootropics. Brain Res Brain Res Rev 1994;19(2):180-222.
3. Kabes J, Sikora J, Pisvejc J, et al. Effect of piracetam on extrapyramidal side effects induced by neuroleptic drugs. Int Pharmacopsychiatry 1982;17(3):185-92.
4. Giurgea C, Salama M. Nootropic Drugs. Prog Neuropsychopharmacol 1977;1:235-247.
5. Pepeu G, Spignoli G. Nootropic drugs and brain cholinergic mechanisms. Prog Neuropsychopharmacol Biol Psychiatry 1989;13(Suppl):S77-88.
6. Pilch H, Muller WE. Piracetam elevates muscarinic cholinergic receptor density in the frontal cortex of aged but not of young mice. Psychopharmacology 1988;94(1):74-8.
7. Tacconi M, Wurtman R. Piracetam: physiological disposition amd mechanism of action. In: Fahn S, editor. Advances in Neurology. NY: Raven Press; 1986.
8. Sikora J, Kabes J, Pisvejc J. [Management of neuroleptic side-effects with piracetam (author's transl)]. Cesk Psychiatr 1981;77(2):137-42.
9. Kabes J, Sikora J, Stary O, et al. [Effectiveness of piracetam in tardive dyskinesia - double-blind cross-over controlled trial with a placebo]. Cesk Psychiatr 1983;79(5):339-45.
10. Chaturvedi SK. Piracetam for drug-induced dyskinesia. J Clin Psychiatry 1987;48(6):255.
11. Obeso JA, Artieda J, Quinn N, et al. Piracetam in the treatment of different types of myoclonus. Clin Neuropharmacol 1988;11(6):529-36.
12. Piperidou C, Maltezos E, Kafalis G, et al. Piracetam for choreoathetosis. Lancet 1988;2(8616):906.
13. Fleischhacker WW, Roth SD, Kane JM. The pharmacologic treatment of neuroleptic-induced akathisia. J Clin Psychopharmacol 1990;10(1):12-21.
14. Fehr C, Dahmen N, Klawe C, et al. Piracetam in the treatment of tardive dyskinesia and akathisia: a case report. J Clin Psychopharmacol 2001;21(2):248-9.
15. Chouinard G, Ross-Chouinard A, Annable L, Jones B. Extrapyramidal Symptom Rating Scale. Can J Neurol Sci (abstract) 1980;7:233.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75
* DSM-IV diagnosis of tardive dyskinesia
* stable psychotropic regimen of a month prior to entry
* duration of TD for at least one year
* hospitalization at our Center

Exclusion Criteria:

* family history of Huntington's disease
* drug or alcohol abuse
* concurrent medial illness or neurological disorder that may have contributed to the diagnosis of TD

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-08

PRIMARY OUTCOMES:
Extrapyramidal Symptom Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lerner, MD, PhD, Principal Investigator — Ben-Gurion University of the Negev; Igor Libov, MD, Principal Investigator — Beersheva Mental Health Center
Locations (1):
- Beersheva Mental Health Center, Beersheva, Israel

REFERENCES:
- [Derived] Libov I, Miodownik C, Bersudsky Y, Dwolatzky T, Lerner V. Efficacy of piracetam in the treatment of tardive dyskinesia in schizophrenic patients: a randomized, double-blind, placebo-controlled crossover study. J Clin Psychiatry. 2007 Jul;68(7):1031-7. doi: 10.4088/jcp.v68n0709. PMID 17685739